CLINICAL TRIAL: NCT00252252
Title: Crossover Trial of VPAP (Variable Positive Airway Pressure) Ventilation Versus AutoVPAP in Neuromuscular and Chest Wall Disease: Effects on Nocturnal Hypoventilation, Sleep Quality and Tolerance
Brief Title: AutoVPAP Versus VPAP; Assessment of Sleep and Ventilation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ResMed (Industry)
Collaborators: Royal Brompton & Harefield NHS Foundation Trust (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2005LF009B; REC Ref No 05/Q0404/001
Record Dates: First submitted 2005-11-09; First posted 2005-11-11 (Estimated); Last update posted 2008-06-24 (Estimated); Status verified 2008-06

CONDITIONS: Chest Wall Disorder; Neuromuscular Disease
MeSH Terms: conditions — Neuromuscular Diseases

INTERVENTIONS:
Device: VPAP non-invasive ventilator
Device: AutoVPAP non-invasive ventilator

SUMMARY:
The aim of the study is to compare the effects of a modified form (AutoVPAP) of the VPAP non-invasive ventilator versus standard VPAP ventilation on sleep quality and breathing during sleep in stable patients with nocturnal hypoventilation due to restrictive ventilatory disorders (eg. neuromuscular disease or chest wall disorder).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-80 years
* Nocturnal hypoventilation (nocturnal peak transcutaneous PCO2 > 6.5 kPa when breathing spontaneously) with
* Congenital neuromuscular disease (eg. Duchenne muscular dystrophy, congenital muscular dystrophy), acquired neuromuscular disease (eg. old polio, bilateral diaphragm paralysis) or chest wall disease (eg. idiopathic scoliosis, thoracoplasty)
* Recruited from 1300 patients attending Royal Brompton Hospital Lind ward ventilator clinic.
* All patients will be familiar with non-invasive ventilation use but currently using a ventilator which is not a VPAP model eg. BiPAP Harmony, Breas PV403.
* Able to understand treatment and protocol

Exclusion Criteria:

* Unstable respiratory failure (PaO2 < 7.5 kPa, PaCO2 > 8.0 kPa,
* Uncontrolled heart failure or arrhythmia
* Moderate or severe bulbar weakness.
* Unable to understand treatment or protocol

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2005-11; Primary Completion 2007-06 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Compare objective measures of sleep, sleep related ventilation and daytime respiratory function between the two treatment devices, VPAP and AutoVPAP.

SECONDARY OUTCOMES:
Compare tolerance of AutoVPAP versus standard VPAP
Compare effects on overnight heart rate variation (as a measure of autonomic stress)
Measure of hours of use of device
Measure of effect on daytime sleepiness

CONTACTS AND LOCATIONS:
Overall Officials: Anita Simonds, MD, FRCP, Principal Investigator — Royal Brompton & Harefield NHS Foundation Trust
Locations (1):
- Royal Brompton Hospital, London, Greater London, United Kingdom

REFERENCES:
- [Derived] Jaye J, Chatwin M, Dayer M, Morrell MJ, Simonds AK. Autotitrating versus standard noninvasive ventilation: a randomised crossover trial. Eur Respir J. 2009 Mar;33(3):566-71. doi: 10.1183/09031936.00065008. PMID 19251798